CLINICAL TRIAL: NCT01679392
Title: Transversus Abdominis Plane Block: A Placebo-controlled Study in Healthy Volunteers
Brief Title: A Study Investigating Properties of the Transversus Abdominis Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillerod Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Kai Henrik Wiborg Lange, Associate Professor, Hillerod Hospital, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-1-2011-030; 2011-004719-22 (EudraCT Number)
Record Dates: First submitted 2012-08-27; First posted 2012-09-06 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Anesthesia, Local
Keywords: Transversus abdominis plane block; Ultrasound guided nerve block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ropivacaine (Experimental): Unilateral transversus abdominis plane block with 20 ml ropivacaine (7.5 mg/ml)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Unilateral, single shot, ultrasound-guided, transversus abdominis plane block with 20 ml ropivacaine (7.5 mg/ml)
  Other Names: Naropin

SUMMARY:
In this study we investigate the following properties of the transversus abdominis plane block in healthy volunteers:

1. Cutaneous analgesic distribution
2. Muscular affection
3. Reproducibility

ELIGIBILITY:
Inclusion Criteria:

* Capable
* American society of anesthesiologists classification 1 or 2
* Written informed consent

Exclusion Criteria:

* Age below 18 years
* American society of anesthesiologists classification above 2
* Body weight below 50 kg
* Body mass index > 35 kg/m2
* Previous abdominal surgery
* Acute or chronic pain
* Use of pain medication less than 24 h prior to study start
* Allergy to local anesthetics
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Cutaneous analgesic distribution | 90 min
  Cutaneous analgesic distribution 90 min after transversus abdominis plane block administration

SECONDARY OUTCOMES:
Muscular affection of the transversus abdominis plane block | 90 min
  Abdominal wall muscle affection of the transversus abdominal plane block measured by ultrasonography under standardized conditions
Reproducibility of the transversus abdominis plane block | At least 2 days
  Reproducibility of the transversus abdominis plane block with respect to:
  1. Cutaneous analgesic distribution
  2. Abdominal wall muscle affection measured in the same individual separated by at least 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Kion Bo Støving, MD, Principal Investigator — Hillerod Hospital, Denmark; Charlotte Rosenstock, MD, Study Director — Hillerod Hospital, Denmark; Kai Lange, MD, Study Director — Hillerod Hospital, Denmark
Locations (1):
- Hillerød Hospital, Hillerød, Denmark